CLINICAL TRIAL: NCT06044961
Title: Radiomics-based Models for the Prediction of Pathological Response to Neoadjuvant Therapy in Gastric and Gastroesophageal Cancer
Acronym: RADI-S
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Agnes Annamaria, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5297
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Patients With Locally Advanced Carcinoma of the Stomach and Oesophagogastric Junction
Keywords: stomach cancer; esophagogastric junction.; locally advanced carcinoma of the stomach; radiomics
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: CT scan — All pre-operative CT scan collected

SUMMARY:
Identifying predictors of response to neoadjuvant therapy in gastric and gastro-oesophageal cancer early in the history of the disease would ensure optimal treatment planning.

The study aims to apply radiomics for the prediction of response to neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced stomach cancer undergoing neoadjuvant chemotherapy and gastrectomy between January 2005 and August 2022

Exclusion Criteria:

* Siewert 1 tumors;
* Patients who have received neoadjuvant with the addition of a biological drug;
* Patients who have received radiotherapy;
* Patients without staging CT scan or with insufficient image quality in terms of phases performed, pixel spacing, slide thickness (mandatorily: > 5 mm) or artefacts.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locally advanced stomach cancer
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-01-01; Primary Completion 2022-08-30 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Use of radiomics | 1 month
  Apply radiomics for predicting response to neoadjuvant therapy.